CLINICAL TRIAL: NCT04165187
Title: The Effects of Body Awareness Therapy on Pain, Balance and Functional Capacity in Patients With Knee Osteoarthritis
Brief Title: Effects of Body Awareness Therapy in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Kübra Alpay, Lecturer of Pysiotherapy and Rehabilitation Department, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kubra1
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; body awareness therapy; pain; functional capacity
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAT+Home exercise program (Experimental): The patients in this group will participate in BAT for 3 days a week for 6 weeks in addition to home exercise program.
  Interventions: Other: Body Awareness Therapy; Other: Home exercise program
- Home exercise program (Active Comparator): The patients in the control group will perform home exercise program, two times a day, 7 days a week for 6 weeks.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Body Awareness Therapy — Body scanning, stretch-release movements, centralization, contact with the ground, postural stability, movement flow and free breathing will be performed during sessions in lying, sitting and standing positions.
  Arms: BAT+Home exercise program
Other: Home exercise program — Home exercise program will consist of joint range of motion, stretching, strengthening and proprioceptive exercises for lower extremity.

SUMMARY:
The aim of this study is to investigate the effect of Body Awareness Therapy (BAT) on pain, balance and functional capacity in patients with knee osteoarthritis.

Individuals will divided into two groups: training group and control group. Both groups will receive exercise training as a home program. Individuals in study group will participate in BAT training 3 days for 6 weeks. Assessments will be made before and after the 6-week study program.

DETAILED DESCRIPTION:
Symptoms such as pain, morning stiffness, and decreased muscle strength lead to a decrease in functional capacity and quality of life in knee osteoarthritis. It is estimated that 80% of patients with osteoarthritis have movement limitation and 25% are unable to perform significant daily activities. It is also stated that increases the risk of falls due to decrease proprioception in patients with knee osteoarthritis. In addition to physical symptoms, it is reported in the literature that symptoms such as sleep disturbance, depression and anxiety are seen and play a role in pain experience.

It is stated in the literature that hypersensitivity of the central nervous system causes painful perception of normal body functions in chronic osteoarthritis, which leads patients to compensatory and dysfunctional movement strategies.

Body Awareness Therapy (BAT) is a mind-body treatment approach directed towards awareness of body senses and how the body is used. The aim is to integrate the body and soul in the individual's experiences and to restructure body awareness and control.

The aim of this study is to investigate the effect of BAT on pain, balance and functional capacity in patients with knee osteoarthritis.

The study will consist of patients with stage 2-3 knee osteoarthritis according to Kellgren-Lawrence classification.

The individuals included in the study will be divided into two groups as training and control groups using a computer-based randomization program.

Both groups will be given a home program consisting of joint range of motion, stretching, strengthening and proprioceptive exercises. The control group will perform home exercise program and follow up will be made at once a week. The training group will participate in BAT for 3 days/week for 6 weeks in addition to home exercise program. Assessments will be made before and after the 6-week study program.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee Osteoarthritis
* Stage 2 -3 according to Kellgren - Lawrence Classification

Exclusion Criteria:

* Previous surgery in the lower extremity
* Neuromuscular disease
* Vestibular pathology
* Physiotherapy intervention or intra-articular injection within the last 6 months

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | six weeks
  change in knee pain intensity from baseline at 6 weeks,"0" point means that there is no pain, "10" point indicates severity of pain
Single leg stability | six weeks
  change in overall stability index of athlete single leg stability test in Biodex Balance System (BBS) from baseline at 6 weeks. Stability level of platform will be set as static. The results can be compared with normative values in the BBS. Lower scores indicate better stability and higher scores mean poor balance.
6 minute walk test | six weeks
  change in walking distance from baseline at 6 weeks
5 times sit to stand test | six weeks
  change in time needed to complete the test from baseline at 6 weeks
Stair climb test | six weeks
  change in time needed to complete the test form baseline at 6 weeks
Hand-held dynamometer | six weeks
  changes quadriceps muscle strength from baseline at 6 weeks

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities osteoarthritis index (WOMAC) | six weeks
  change in scores from baseline at 6 weeks. Index consists of 24 items. In index maximum score is 96 points and minimum score is 0 point. Higher scores indicate worse symptoms, physical limitation.
Fall risk | six weeks
  change in overall stability index of fall risk test in Biodex Balance System from baseline at 6 weeks. Lower scores indicate better balance and high scores mean high risk for fall.
joint range of motion | six weeks
  change in knee joint range of motion from baseline at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Alpay, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Eyup, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alpay K, Sahin M. Effects of basic body awareness therapy on pain, balance, muscle strength and functionality in knee osteoarthritis: a randomised preliminary trial. Disabil Rehabil. 2023 Dec;45(26):4373-4380. doi: 10.1080/09638288.2022.2151650. Epub 2022 Nov 29. PMID 36444879